CLINICAL TRIAL: NCT04862143
Title: Open-label, Multicenter, Pilot-trial Evaluating the Safety and Utility of a Hybrid Decentralized Clinical Trial (DCT) Approach Using a TELEmedicine Platform in Patients With HR-positive/HER2-negative Advanced Breast Cancer With a PIK3CA Mutation Treated With Alpelisib - Fulvestrant TELEPIK Trial
Brief Title: Pilot Decentralized Clinical Trial in Men and Pre and Post-menopausal Women With Breast Cancer and a Specific Mutation (PIK3CA) Treated With Alpelisib in Combination With Fulvestrant
Acronym: TELEPIK
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study early terminated due to low enrollment compared to the anticipated figures
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719A03201; 2020-005882-15 (EudraCT Number)
Record Dates: First submitted 2021-04-21; First posted 2021-04-27 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Advanced Breast Cancer
Keywords: Decentralized clinical trial; advanced breast cancer; PIK3CA mutation; alpelisib
MeSH Terms: interventions — Alpelisib; Fulvestrant; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alpelisib + fulvestrant (Experimental): Participants were administered alpelisib at a daily dose of 300 mg for 12 cycles of 28 days and fulvestrant at a dose of 500 mg via intramuscular injection on Cycle 1 Day 1 and Cycle 1 Day 15, and Day 1 of each subsequent cycle up to Cycle 12. Pre-menopausal women also received goserelin at a dose of 3.6 mg on Day 1 of each cycle.
  Interventions: Drug: Alpelisib; Drug: Fulvestrant; Drug: Goserelin

INTERVENTIONS:
Drug: Alpelisib — Participants received a daily oral dose of 300 mg of alpelisib film-coated tablets for a total of 12 cycles, with each cycle lasting 28 days.
  Other Names: BYL719
Drug: Fulvestrant — Participants were administered fulvestrant at a dose of 500 mg via intramuscular injection on Cycle 1 Day 1 and Cycle 1 Day 15, and on Day 1 of each 28-day cycle thereafter until Cycle 12.
Drug: Goserelin — Pre-menopausal women were administered a dose of 3.6 mg of goserelin injection via intramuscular route, beginning on Cycle 1 Day 1. Subsequently, the same dose was administered on Day 1 of each 28-day cycle throughout the study.

SUMMARY:
The study was designed to identify and register practical observations and experiences in connection with planning and implementing decentralized, patient-centered clinical trials at a geographic distance with virtual elements.

DETAILED DESCRIPTION:
The purpose of this open-label, single arm, multi-center, Phase II interventional pilot trial was to evaluate if a decentralized clinical trial (DCT) using a telemedicine platform offers a satisfactory, safe and suitable management for HR-positive/HER2-negative participants with advanced breast cancer harboring a PIK3CA mutation and treated with alpelisib plus fulvestrant. The trial utilized a hybrid DCT approach to reduce participant burden by bringing visits, services, and supplies closer to them.

The planned duration of treatment was 12 cycles of 28 days. Participants could discontinue treatment earlier due to unacceptable toxicity, disease progression and/or decision made at the discretion of the investigator or the participant.

On-site visits occurred during screening, at Cycle 1 Day 1 (baseline), and at end-of-trial. Visits at the local oncologist practice were planned on Day 1 of Cycle 2, Cycle 4, Cycle 7, and Cycle 10. Other visits were performed by a district nurse, either at home or at the local oncologist's practice, depending on the participant's preference.

During the on-site visit on Cycle 1, Day 1, participants were trained on using the telemedicine platform, and other monitoring devices used during remote participation: a glucometer and a smartphone with the telemedicine application installed. Study treatment was also initiated during this visit. The participants were then transitioned to remote participation enabled by the telemedicine platform with support of local healthcare providers (local oncologist, district nurse, or other qualified healthcare professional) under the investigator's oversight.

Discontinuation of remote participation was not a reason for trial termination. Participants who did not wish to continue with remote participation had the option to attend on-site visits.

The study planned to enroll approximately 20 participants, however the study was terminated prematurely with only 2 participants enrolled. The decision to terminate the study was due to delays during the start-up period and due to low enrollment. The decision to terminate was not related to any potential safety concern with alpelisib.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant is an adult ≥18 years old at the time of consent
2. Participant with ABC (loco regionally recurrent or metastatic) not amenable to curative therapy.
3. Participant with a histologically and/or cytologically confirmed diagnosis of ER-positive and/or PR-positive breast cancer by local laboratory.
4. Participant with a confirmed HER2-negative ABC.
5. Participant with a pathology report confirming PIK3CA mutant status by a certified laboratory using a validated PIK3CA mutation assay (from either tissue or blood).
6. Participant was willing to operate a smartphone compatible with the software of the medical device and willing to manage applications
7. Participant was willing to use the telemedicine platform and to follow the remote participant monitoring procedure.

Key Exclusion Criteria:

1. Participant had received prior treatment with any PI3K, mTOR or AKT inhibitor.
2. Participant with known hypersensitivity to alpelisib or fulvestrant, or to any of the excipients of alpelisib or fulvestrant.
3. Participant participated in a prior investigational study within 30 days prior to the start of trial treatment or within 5 half-lives of the trial treatment, whichever was longer.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1606

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 1 center from Sweden
Period: Overall Study
Arm/Group | Alpelisib + Fulvestrant
Started | 2
Completed | 0
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Study terminated by sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54 (0)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender details were not collected from any participant
  Participants
    Unknown | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Participant Satisfaction Assessed Through the Trial Feedback Questionnaire (TFQ)
Description: The TFQ was designed to capture the patient's experience during a clinical trial. The questionnaire consisted of 23 questions that assessed various aspects of the trial experience. Each question in the TFQ scored on a scale ranging from 1 (representing the worst response) to 5 (representing the best response). To calculate the total score, the scores obtained from each of the 23 questions were summed up. The resulting sum represented the participant's total score, which could ranged from 23 (indicating the lowest possible score) to 115 (indicating the highest possible score).
Time Frame: Baseline, and on Day 1 of Cycle 4 and 7. Cycle= 28 days
Population: All enrolled participants who received at least one dose of any component of study treatment
Measure: Median (Full Range); unit: Score on a Scale
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 2
Score on a Scale
  Baseline | 99.5 [92 to 107]
  Cycle 4 Day 1: number analyzed (Participants) | 1
  Cycle 4 Day 1 | 89
  Cycle 7 Day 1: number analyzed (Participants) | 1
  Cycle 7 Day 1 | 98

2. Secondary Outcome: Patient Retention on the Decentralized Clinical Trial (DCT) Approach
Description: Patient retention on the DCT approach was calculated as the percentage of participants on remote monitoring for participants still on treatment
Time Frame: At 3 and 6 months
Population: Participants receiving treatment at the specified time points
Measure: Count of Participants; unit: Participants
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 1
Participants
  3 months | 1
  6 months | 1

3. Secondary Outcome: Number of Unscheduled In-clinic Visits
Description: Unscheduled in-clinic visits were defined as visits that were originally intended to be conducted remotely but were ultimately carried out on-site, or visits that were not originally scheduled but took place on-site or at the local oncologist's (regional hospital).
  The total number of unscheduled in-clinic visits was evaluated
Time Frame: From the date of the first study treatment up to the end of study, assessed up to 6 months
Population: All enrolled participants who received at least one dose of any component of study treatment
Measure: Number; unit: Visits
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 2
Visits | 0

4. Secondary Outcome: Number of Unscheduled In-clinic Visits Because of Safety Reasons
Description: Unscheduled in-clinic visits were defined as visits that were originally intended to be conducted remotely but were ultimately carried out on-site, or visits that were not originally scheduled but took place on-site or at the local oncologist's (regional hospital).
  The total number of unscheduled in-clinic visits that were prompted by safety reasons was evaluated
Time Frame: From the date of the first study treatment up to the end of study, assessed up to 6 months
Population: All enrolled participants who received at least one dose of any component of study treatment
Measure: Median (Full Range); unit: Visits
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 2
Visits | 0 [0 to 0]

5. Secondary Outcome: Number of Unscheduled In-clinic Visits Per Participant in the Study
Description: Unscheduled in-clinic visits were defined as visits that were originally intended to be conducted remotely but were ultimately carried out on-site, or visits that were not originally scheduled but took place on-site or at the local oncologist's (regional hospital).
  The total number of unscheduled in-clinic visits per participants was evaluated
Time Frame: From the date of the first study treatment up to the end of study, assessed up to 6 months
Population: All enrolled participants who received at least one dose of any component of study treatment
Measure: Median (Full Range); unit: Visits per participant
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 2
Visits per participant | 0 [0 to 0]

6. Secondary Outcome: Number of Participants Who Discontinue Treatment Due to Adverse Events (AEs)
Description: An AE refers to any untoward medical occurrence, such as an unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease.
  The number of participants who discontinued the treatment due to adverse events was evaluated
Time Frame: From the date of the first study treatment up to the end of treatment, assessed up to 6 months
Population: All enrolled participants who received at least one dose of any component of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 2
Participants | 1

7. Secondary Outcome: Number of Participants With Dose Reductions/Interruptions for Alpelisib
Description: Number of participants with dose reductions and interruptions for alpelisib
Time Frame: From the date of the first study treatment up to the end of treatment, assessed up to 6 months
Population: All enrolled participants who received at least one dose of any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 2
Participants
  Dose interruptions | 1
  Dose reductions | 1

8. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)- Hyperglycemia, Rash and Diarrhea
Description: AESIs (Adverse Events of Special Interest) are defined as events, whether serious or non-serious, that are of scientific and medical concern specific to the sponsor's product or program. These events may require ongoing monitoring and communication by the investigator to the sponsor. For this study, the following AESIs were defined: hyperglycemia, rash, and diarrhea.
  The number of participants experiencing these events per the Common Terminology Criteria for Adverse Events (CTCAE) v4.03 was evaluated.
Time Frame: From the date of the first study treatment up to the end of study, assessed up to 6 months
Population: All enrolled participants who received at least one dose of any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 2
Participants
  Diarrhea | 1
  Hyperglycaemia | 2
  Rash | 0

9. Secondary Outcome: Number of Participants With Adverse Events (AEs) Leading to In-clinic Visits
Description: An AE refers to any untoward medical occurrence, such as an unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease.
  The number of participants with AEs per the Common Terminology Criteria for Adverse Events (CTCAE) v4.03 leading to in-clinic visits was assessed.
Time Frame: From the date of the first study treatment up to the end of study, assessed up to 6 months
Population: All enrolled participants who received at least one dose of any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 2
Participants | 0

10. Secondary Outcome: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 questionnaire contained 30 items and was composed of both multi-item scales and single item measures. These included five functional scales (physical, role, emotional, cognitive, and social functioning), three symptom scales (fatigue, nausea/vomiting, and pain), six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial impact), and a global health status/quality of life (QoL) scale.
  All of the scales and single items ranged from 0 to 100. A high scale score represented a higher response level. Thus, a high score for a functional scale indicated a high/healthy level of functioning, a high score for the QoL indicated high QoL, but a high score for a symptom scale/single item indicated a high level of symptomatology/problems.
  The EORTC QLQ-C30 scores for all functional and symptom scales were evaluated
Time Frame: Baseline, and on Day 1 of Cycle 4, and 7 and end of treatment, assessed up to 6 months. Cycle= 28 days
Population: All enrolled participants who received at least one dose of any study treatment. Number analyzed indicates the number of participants with data available at the designated time point.
Measure: Median (Full Range); unit: Score on a Scale
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 2
Score on a Scale
  QoL- Baseline | 75 [67 to 83]
  QoL- Cycle 4 Day 1: number analyzed (Participants) | 1
  QoL- Cycle 4 Day 1 | 83
  QoL- Cycle 7 Day 1: number analyzed (Participants) | 1
  QoL- Cycle 7 Day 1 | 92
  QoL- End of Treatment | 75 [67 to 83]
  Physical Functioning- Baseline | 90 [80 to 100]
  Physical Functioning- Cycle 4 Day 1: number analyzed (Participants) | 1
  Physical Functioning- Cycle 4 Day 1 | 93
  Physical Functioning- Cycle 7 Day 1: number analyzed (Participants) | 1
  Physical Functioning- Cycle 7 Day 1 | 100
  Physical Functioning-End of Treatment | 86.5 [80 to 93]
  Role Functioning- Baseline | 91.5 [83 to 100]
  Role Functioning- Cycle 4 Day 1: number analyzed (Participants) | 1
  Role Functioning- Cycle 4 Day 1 | 100
  Role Functioning- Cycle 7 Day 1: number analyzed (Participants) | 1
  Role Functioning- Cycle 7 Day 1 | 100
  Role Functioning-End of Treatment | 83.5 [67 to 100]
  Emotional Functioning- Baseline | 71 [67 to 75]
  Emotional Functioning- Cycle 4 Day 1: number analyzed (Participants) | 1
  Emotional Functioning- Cycle 4 Day 1 | 83
  Emotional Functioning- Cycle 7 Day 1: number analyzed (Participants) | 1
  Emotional Functioning- Cycle 7 Day 1 | 92
  Emotional Functioning- End of treatment | 83 [83 to 83]
  Cognitive Functioning- Baseline | 91.5 [83 to 100]
  Cognitive Functioning- Cycle 4 Day 1: number analyzed (Participants) | 1
  Cognitive Functioning- Cycle 4 Day 1 | 100
  Cognitive Functioning- Cycle 7 Day 1: number analyzed (Participants) | 1
  Cognitive Functioning- Cycle 7 Day 1 | 100
  Cognitive Functioning- End of treatment | 75 [67 to 83]
  Social Functioning- Baseline | 91.5 [83 to 100]
  Social Functioning- Cycle 4 Day 1: number analyzed (Participants) | 1
  Social Functioning- Cycle 4 Day 1 | 100
  Social Functioning- Cycle 7 Day 1: number analyzed (Participants) | 1
  Social Functioning- Cycle 7 Day 1 | 100
  Social Functioning- End of treatment | 91.5 [83 to 100]
  Fatigue- Baseline | 22 [0 to 44]
  Fatigue- Cycle 4 Day 1: number analyzed (Participants) | 1
  Fatigue- Cycle 4 Day 1 | 22
  Fatigue- Cycle 7 Day 1: number analyzed (Participants) | 1
  Fatigue- Cycle 7 Day 1 | 0
  Fatigue- End of treatment | 33 [22 to 44]
  Nausea/vomiting- Baseline | 0 [0 to 0]
  Nausea/vomiting- Cycle 4 Day 1: number analyzed (Participants) | 1
  Nausea/vomiting- Cycle 4 Day 1 | 17
  Nausea/vomiting- Cycle 7 Day 1: number analyzed (Participants) | 1
  Nausea/vomiting- Cycle 7 Day 1 | 0
  Nausea/vomiting- End of treatment | 0 [0 to 0]
  Pain- Baseline | 8.5 [0 to 17]
  Pain- Cycle 4 Day 1: number analyzed (Participants) | 1
  Pain- Cycle 4 Day 1 | 0
  Pain- Cycle 7 Day 1: number analyzed (Participants) | 1
  Pain- Cycle 7 Day 1 | 0
  Pain- End of treatment | 16.5 [0 to 33]

11. Secondary Outcome: EuroQol 5-Dimension 5-Level (EQ-5D-5L)- Visual Analog Scale (VAS) Score
Description: The 5-level EQ-5D (EQ-5D-5L) questionnaire is a standardized measure of health status. The EQ-5D descriptive system comprises of the 5 following dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Along with the five dimensions of health, the EQ-5D-5L includes a VAS where respondents rate their overall health status on a scale from 0 to 100, where 0 represents the worst possible health state and 100 represents the best possible health state.
  The EQ-5D-5L VAS scores were evaluated
Time Frame: Baseline, and on Day 1 of Cycle 4, and 7 and end of treatment, assessed up to 6 months. Cycle= 28 days
Population: as for outcome 10
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 2
Score on a scale
  Baseline | 80 [75 to 85]
  Cycle 4 Day 1: number analyzed (Participants) | 1
  Cycle 4 Day 1 | 93
  Cycle 7 Day 1: number analyzed (Participants) | 1
  Cycle 7 Day 1 | 95
  End of treatment | 82.5 [70 to 95]

12. Secondary Outcome: Brief Pain Inventory Short Form (BPI-SF) Scores
Description: The BPI-SF was a questionnaire used to assess pain intensity and interference with daily activities. The Pain Severity Subscale included four questions asking individuals to rate their pain intensity on a scale from 0 to 10, with higher scores indicating more severe pain. The Pain Interference Subscale consisted of seven items that assessed how pain had interfered with activities, rated on the same scale. Both subscales had a total score range of 0 to 10, with higher scores indicating more significant pain or interference.
Time Frame: Baseline, and on Day 1 of Cycle 4, and 7 and end of treatment, assessed up to 6 months. Cycle= 28 days
Population: as for outcome 10
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 2
Score on a scale
  Pain severity- Baseline | 1.63 [1.25 to 2.00]
  Pain severity- Cycle 4 Day 1: number analyzed (Participants) | 1
  Pain severity- Cycle 4 Day 1 | 0
  Pain severity- Cycle 7 Day 1: number analyzed (Participants) | 1
  Pain severity- Cycle 7 Day 1 | 0.75
  Pain severity- End of treatment | 1.13 [0.00 to 2.25]
  Pain interference- Baseline | 0.79 [0.00 to 1.57]
  Pain interference- Cycle 4 Day 1: number analyzed (Participants) | 1
  Pain interference- Cycle 4 Day 1 | 0
  Pain interference- Cycle 7 Day 1: number analyzed (Participants) | 1
  Pain interference- Cycle 7 Day 1 | 0
  Pain interference- End of treatment | 1.07 [0 to 2.14]

13. Secondary Outcome: Number of Participants With Progression-free Survival (PFS) According to RECIST 1.1
Description: The number of participants with PFS was defined as the count of participants who did not experience disease progression or death due to any cause during the study. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 based on local radiology review.
Time Frame: Up to 6 months
Population: All enrolled participants who received at least one dose of any component of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: From start up to end of study, assessed up to 6 months
Arm/Group | Alpelisib + Fulvestrant
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alpelisib + Fulvestrant (N=2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Fatigue (General disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Weight decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT04862143/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT04862143/SAP_001.pdf